CLINICAL TRIAL: NCT01978262
Title: A Pilot Study of the Immune Response to Influenza Vaccination and Effect on Reproductive Hormones
Brief Title: Immune and Hormone Response to Influenza Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIR 292; 200-2012-53664-002 (Other Grant/Funding Number: CDC)
Record Dates: First submitted 2013-10-24; First posted 2013-11-07 (Estimated); Results first posted 2018-10-11 (Actual); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Healthy
Keywords: influenza vaccine; cytokines; hormones; progesterone
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- healthy woman (Other): All women are to receive the quadrivalent influenza vaccine
  Interventions: Biological: Seasonal Inactivated Influenza Vaccine

INTERVENTIONS:
Biological: Seasonal Inactivated Influenza Vaccine — Quadrivalent seasonal inactivated influenza vaccine, 0.5 mL intramuscularly
  Other Names: FluZone

SUMMARY:
The purpose of this pilot research project is to look at the effect of the inactivated influenza vaccine (seasonal flu shot) on early signs of immune or germ-fighting response known as cytokines or signal molecules. The investigators also want to see if the timing of vaccine administration has any effect on women's reproductive hormones. The investigators hypothesis is that influenza vaccine given right before ovulation may change the hormone levels usually seen after ovulation. Thi

DETAILED DESCRIPTION:
This study is an open-label, longitudinal study of healthy young women of reproductive age, not on hormonal contraception who receive seasonal inactivated influenza vaccine (IIV). The women will be followed for one menstrual cycle to measure luteinizing hormone surge, estradiol, and progesterone, and then vaccinated with the seasonal inactivated influenza vaccine prior to ovulation during a second month. At the investigator's discretion, or if there is active circulation of influenza virus in Baltimore, the investigators will vaccinate during the first menstrual cycle (prior to ovulation) and then follow for a second menstrual cycle for comparison. After vaccination, they will be followed for cytokine and chemokine responses as well as changes in the concentrations of steroid hormones. This study will evaluate the effect of IIV on inflammatory cytokines and hormonal responses before and after ovulation. Each woman will have 13 visits in addition to a screening visit, and will be followed for 2 complete menstrual cycles.

ELIGIBILITY:
Inclusion Criteria:

* Women 18-39 years of age who are in good health.
* Good general health as a result of review of medical history and/or clinical testing at the time of screening.
* Available for the duration of the trial.
* Willingness to participate in the study as evidenced by signing the informed consent document.
* Willing to be abstinent or to use non-hormonal methods of contraception for the duration of the study.
* History of normal menstrual cycles (26-35 days in length) for at least 3 months.
* Willingness to refrain from routine vaccination (except as administered during study) for the duration of the study.

Exclusion Criteria:

* Use of contraceptive pills, patch, injection or other hormonal therapies in the preceding 3 months (6 months for DepoProvera)
* A history of hypersensitivity, including anaphylaxis to any of the components of IIV or to eggs.
* Previous receipt of a same season licensed influenza vaccine.
* Pregnancy as determined by a positive urine or serum human choriogonadotropin (β-hCG) test at any point during the study or in the preceding 3 months.
* Currently is lactating or breast-feeding.
* Fewer than 3 normal menstrual cycles since conclusion of last pregnancy or last use of hormonal birth control.
* A history of autoimmune disease, or any other chronic medical condition considered clinically significant by the investigator.
* History of HIV, Hepatitis C or active Hepatitis B.
* Known immunodeficiency syndrome.
* History of Guillain-Barré syndrome.
* Use of chronic oral or intravenous administration (≥14 days) of immunosuppressive doses of steroids, i.e., prednisone >10 mg per day, immunosuppressants or other immune-modifying drugs within 30 days of starting this study. (Use of topical, nasal or inhaled steroids is permitted)
* Receipt of a live vaccine within 4 weeks or a killed vaccine within 2 weeks prior to study start or during study.
* Receipt of blood or blood-derived products (including immunoglobulin) within 6 months prior to study vaccination.
* Receipt of another investigational vaccine or drug within 30 days prior to study start, or during study.
* Ongoing, daily use of analgesics or anti-inflammatory medications, including nonsteroidal anti-inflammatories. Occasional use, and use associated with menstrual periods is acceptable.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2013-10; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kawsar R Talaat, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Karen Broder, M.D., Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- Center for Immunization Research; Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

REFERENCES:
- See also: Click here for information about enrolling in this study — http://hopkinsprojectsave.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 103 adult female subjects enrolled and 92 completed study over 3 vaccination seasons from 2013-2017. Each participant served as her own control and followed for 2 months: an Inactivated influenza vaccination (IIV) month and a observation/comparator month.
Pre-assignment Details: Study specific screening occurred prior to enrollment. 180 screens completed
Groups:
- Healthy Women: All women are to receive the quadrivalent influenza vaccine
  Seasonal Inactivated Influenza Vaccine: Quadrivalent seasonal inactivated influenza vaccine, 0.5 mL intramuscularly
Period: Overall Study
Arm/Group | Healthy Women
Started | 103
Completed | 92
Not Completed | 11
Not completed — Withdrawal by Subject | 9
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Women
Number analyzed (Participants) | 92
Age, Continuous [Median (Full Range); unit: years] | 28 [19 to 39.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 86
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 11
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 54
  White | 23
  More than one race | 2
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 92

OUTCOME MEASURES:

1. Primary Outcome: Change in Levels of Progesterone After Influenza Vaccination
Description: To explore whether receipt of IIV during the second week of the menstrual cycle (i.e., the week prior to ovulation) is associated with changes in steroid hormone levels, particularly decreases in progesterone, following ovulation.
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Healthy Women (Vaccine): All women are to receive the quadrivalent influenza vaccine
  Seasonal Inactivated Influenza Vaccine: Quadrivalent seasonal inactivated influenza vaccine, 0.5 mL intramuscularly
- Healthy Women (Comparator): All women are to receive the quadrivalent influenza vaccine
  Seasonal Inactivated Influenza Vaccine: Quadrivalent seasonal inactivated influenza vaccine, 0.5 mL intramuscularly
  Comparator Month
Arm/Group | Healthy Women (Vaccine) | Healthy Women (Comparator)
Number analyzed (Participants) | 92 | 92
ng/ml
  Progesterone Day 0 | 0.62 (1.60) | 0.43 (0.80)
  Progesterone Day 11 | 0.73 (1.40) | 0.59 (0.92)
  Progesterone Day 17 | 4.59 (4.42) | 4.53 (4.13)
  Progesterone Day 21 | 6.72 (4.59) | 6.32 (3.70)
  Progesterone Day 28 | 0.55 (1.03) | 0.92 (1.98)

2. Other Pre Specified Outcome: Cytokine Effect on Reproductive Hormone Levels
Description: To explore whether inflammatory cytokine responses to IIV receipt are associated with changes in reproductive and stress hormone levels.
Time Frame: 2 months
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Cytokine Responses to Influenza Vaccine
Description: Identify optimal biomarkers of the inflammatory response after vaccination.
Time Frame: 2 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 7 days after vaccination, up to 2 months
Arm/Group | Healthy Women
All-Cause Mortality (participants affected / at risk) | 0/92
Serious Adverse Events (participants affected / at risk) | 0/92
Other Adverse Events (participants affected / at risk) | 73/92
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Women (N=92)
Chills (Immune system disorders) | 2 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 (2)
Eythema (Skin and subcutaneous tissue disorders) | 9 (9)
Headache (Immune system disorders) | 23 (31)
Induration (Skin and subcutaneous tissue disorders) | 9 (9)
Malaise (Immune system disorders) | 11 (11)
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (10)
Pain (Skin and subcutaneous tissue disorders) | 62 (72)
Pruritis (Skin and subcutaneous tissue disorders) | 2 (2)
Swelling (Skin and subcutaneous tissue disorders) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-01-24): https://cdn.clinicaltrials.gov/large-docs/62/NCT01978262/SAP_000.pdf
  • Study Protocol (2018-01-24): https://cdn.clinicaltrials.gov/large-docs/62/NCT01978262/Prot_001.pdf